CLINICAL TRIAL: NCT01969110
Title: Additional Effects of Perioperative Immunonutrition on Th1/Th2 Differentiation in Patients Undergoing Pancreaticoduodenectomy
Brief Title: Additional Effects of Perioperative Immunonutrition in Patients Undergoing Pancreaticoduodenectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Katsunori Furukawa, MD, PhD, Chiba University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AEPIPD
Record Dates: First submitted 2013-10-05; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Pancreatic Tumor; Bile Duct Tumor
Keywords: Immunonutrition
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perioperative (Active Comparator): Oral IMPACT (1 L/day) for 5 days before surgery and by enteral feeding after surgery
  Interventions: Dietary Supplement: Oral IMPACT
- Preoperative (Active Comparator): Oral IMPACT 1000ml/day for 5 days (1 L/day) before surgery
  Interventions: Dietary Supplement: Oral IMPACT

INTERVENTIONS:
Dietary Supplement: Oral IMPACT — Oral IMPACT enriched with arginine, omega-3 fatty acids, and RNA by enteral feeding after surgery
  Other Names: Oral IMPACT; Ajinomoto Pharma Co., Ltd, Tokyo, Japan

SUMMARY:
The purpose of this study is to investigate whether perioperative immunonutrition has additional effects on cell-mediated immunity in patients undergoing pancreaticoduodenectomy.

DETAILED DESCRIPTION:
The investigators reported that perioperative immunonutrition had no additional effects compared with preoperative immunonutrition in patients underwent colorectal surgery (Braga M, Gianotti L, Vignali A, Carlo VD. Preoperative oral arginine and n-3 fatty acid supplementation improves the immunometabolic host response and outcome after colorectal resection for cancer. Surgery. 2002; 132:805-14, PMID: 12464864). Object of this study is to investigate the additional effects of perioperative immunonutrition on cell-mediated immunity and incidence of infectious complication after pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing pancreaticoduodenectomy

Exclusion Criteria:

* age younger than 18 years old
* ongoing infection
* gastrointestinal obstruction
* respiratory dysfunction
* cardiac dysfunction
* hepatic dysfunction
* renal failure
* history of recent immunosuppressive or immunological disease
* preoperative evidence of widespread metastatic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
plasma resolvin E1, cell-mediated immunity | 30 days

SECONDARY OUTCOMES:
infectious complication rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Katsunori Furukawa, MD, Study Director — Chiba University
Locations (1):
- Chiba University Hospital, Chiba, Chiba, Japan